CLINICAL TRIAL: NCT06164860
Title: The Effect of Ketogenic Diet Versus Mediterranean Diet on Clinical and Biochemical Markers of Inflammationand in Patients With Obesity and Psoriatic Arthritis
Brief Title: The Effect of Ketogenic Diet Versus Mediterranean Diet in Patients With Obesity and Psoriatic Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, VAIA LAMBADIARI, Professor of Internal Medicine-Endocrinology, Attikon Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 171/9-4-2020
Record Dates: First submitted 2023-12-02; First posted 2023-12-11 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Obesity and Psoriasis
MeSH Terms: conditions — Obesity; Psoriasis | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Other): started with MD
  Interventions: Other: Meditteranean Diet; Other: Ketogenic Diet
- Group B (Other): started with KD
  Interventions: Other: Meditteranean Diet; Other: Ketogenic Diet

INTERVENTIONS:
Other: Meditteranean Diet — The MD provided 20% proteins, 40% fat and 40% carbohydrates. Each participant received a brochure with a template of a daily five course (breakfast, lunch, dinner and two snacks) diet plan that provided several options for each meal and was advised to use it as a guide for the 8-week period
Other: Ketogenic Diet — The KD provided approximately 34% proteins, 55% fat and 11% carbohydrates. The macronutrient targets were successfully met by replacing breakfast and two daily snacks with specifically selected food products provided by Evivios Med. Lunch and dinner were natural protein-rich dishes. Each participant received accurate teaching and a brochure that incorporated a template of a weekly diet plan from an expert dietitian.

SUMMARY:
The aim of our study is to compare the effectiveness of Mediterranean diet (MD) with the isocaloric Ketogenic diet (KD) on clinical and biochemical markers of inflammation in patients with obesity, psoriasis (PSO) and psoriatic arthritis (PsA).

DETAILED DESCRIPTION:
Overall, twenty patients with body mass index (BMI) >30 kg/m2, PSO and PsA under constant systematic treatment for at least 3 months will be included in the study. They will randomly assign to two groups, starting either with MD or KD for a period of 8 weeks. After a 6-week washout interval, the two groups will cross over to the other type of diet for the same 8-week period. The primary endpoint is the change in Psoriasis Area and Severity Index (PASI) and the Disease Activity Index for Psoriatic Arthritis (DAPSA) score, 8 weeks after each diet intervention. Secondary endpoints are changes in biochemical markers of inflammation (IL-6, IL-17, IL-22, IL-23) , in metabolic and anthropometric parameters.

ELIGIBILITY:
Inclusion Criteria:

1. age above 18 years
2. body mass index (BMI) >30 kg/m2
3. diagnosis of psoriasis and psoriatic arthritis under constant systematic treatment with biologic agents and/or synthetic disease-modifying anti-rheumatic drugs (DMARDs) for at least 3 months.
4. ΔPASI SCORE<75, with moderate or severe activity in joints ( > 3 swollen &> 3 tender joints ή DAPSA< 14).

Exclusion Criteria:

1. participation in another study
2. eGFR<60ml/min/1.73m2
3. malignancy
4. severe hepatic disorder
5. HbA1C>10%
6. use of glucagon-like-petide-1 analogues

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Psoriasis Area and Severity Index score | eight weeks
  The primary endpoint is changes in Psoriasis Area and Severity Index (PASI), 8 weeks after each diet intervention.(score range: 0-72; higher scores indicate more severe disease).
Disease Activity Index for Psoriatic Arthritis score | eight weeks
  The primary endpoint is changes in Disease Activity Index for Psoriatic Arthritis (DAPSA) score, 8 weeks after each diet intervention.(DAPSA<4: remission, DAPSA 4-14: low disease activity, DAPSA:14-28:moderate disease activity, DAPSA>28: high disease activity)

SECONDARY OUTCOMES:
Interleukin-6 | eight weeks
  Secondary endpoints were biochemical markers of inflammation (IL-6) 8 weeks after KD compared to 8-weeks MD diet intervention.
Interleukin-17 | eight weeks
  Secondary endpoints were biochemical markers of inflammation (IL-17) 8 weeks after KD compared to 8-weeks MD diet intervention.
Interleukin-22 | eight weeks
  Secondary endpoints were biochemical markers of inflammation (IL-22) 8 weeks after KD compared to 8-weeks MD diet intervention.
Interleukin-23 | eight weeks
  Secondary endpoints were biochemical markers of inflammation (IL-23) 8 weeks after KD compared to 8-weeks MD diet intervention.
Glucagon Like Peptide-1 | eight weeks
  The investigators assessed changes in Glucagon Like Peptide-1 levels 8-weeks after KD compared to 8-weeks MD diet intervention.
Oxyntomodulin | eight weeks
  The investigators assessed changes in Oxyntomodulin levels 8-weeks after KD compared to 8-weeks MD diet intervention.
Peptide YY | eight weeks
  The investigators assessed changes in Peptide YY levels 8-weeks after KD compared to 8-weeks MD diet intervention.
Ghrelin | eight weeks
  The investigators assessed changes in Ghrelin levels 8-weeks after KD compared to 8-weeks MD diet intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Vaia Lambadiari, Athens, Attica, Greece